CLINICAL TRIAL: NCT01250249
Title: A Randomized, Open Label, Single-period, Single-treatment, Controlled Multi Center Phase Iii Study of Comparing Safety and Reactogenecity of Lyophilized BCG Vaccine ip (0.1 mg in 0.1 ml) of Green Signal Bio Pharma Private Limited India With BCG Vaccine (0.1 mg in 0.1 ml) of Serum Institute of India Limited (SIIL),India in 120 Healthy Children.
Brief Title: A Study of Comparing Safety and Reactogenicity, of Lyophilized BCG Vaccine IP of Green Signal Bio Pharma Private Limited, India With BCG Vaccine of Serum Institute of India Limited in 120 Healthy Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Signal Biopharma Private Limited (Industry)
Responsible Party: Mr.Sajjanadhasan.VJ, Green Signal Biopharma Private Limited
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BCGV/034/08
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: To compare Safety and Reactogenecity of BCG vaccine of Green Signal Biopharma Private Limited with BCG vaccine of serum institute of India limited

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BCG Vaccine - Intradermal injection (Active Comparator): Subjects must be in the age group of 0 - 14 years of age.
  2. Subject's parent should be able to understand and have to sign the informed consent form after being explained by the investigator. They must be aware of the experimental nature of the therapy, its potential benefits, side effects and risks.
  3. Ability to comply with the schedule of treatment and follow-up.
  4. Absence of BCG scar
  5. Tuberculin negative
  6. No evidence of any other infection
  7. No evidence of skin disease
  Skin testing with tuberculin is not generally carried out before giving BCG but when performed, those who are found to be positive reactors need not to be immunized
  Interventions: Biological: BCG Vaccine IP - Serum Institute of India

INTERVENTIONS:
Biological: BCG Vaccine IP - Serum Institute of India — 0.1 ml for adults and children aged 1 month and over 0.05 ml for infants under 1 month of age
  Other Names: BCG Vaccine IP (SIIL)

SUMMARY:
To compare Safety and Reactogenecity of BCG vaccine of Green Signal Biopharma Private Limited India with BCG vaccine of serum institute of India limited (SIIL), India in 120 healthy children.

DETAILED DESCRIPTION:
The study was conducted in the objective to compare the safety and reactogenecity of BCG Vaccine of Green Signal Bio pharma Private Limited India(Test) with BCG vaccine of Serum Institute of India(Reference) in 120 healthy children.

The above study was conducted in multi centers(2 centers - Chennai & Bangalore). The study was conducted as per the protocol approved by DCGI and Madras ethical Committee.

A single dose was administedred to all the subjects and it was inferred that all the 120 subjects vaccinated were safe. Further, the reactogenecity was confirmed after 90th day by PPD administration to all the subjects. Based on the above observations it was well identified that test vaccine can be safely administered to children and it is well tolerated and accepted by the subjects. More over statistically it is inferred that there is no significant variation between the test and reference vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be in the age group of 0 - 14 years of age.
2. Subject's parent should be able to understand and have to sign the informed consent form after being explained by the investigator. They must be aware of the experimental nature of the therapy, its potential benefits, side effects and risks.
3. Ability to comply with the schedule of treatment and follow-up.
4. Absence of BCG scar
5. Tuberculin negative
6. No evidence of any other infection
7. No evidence of skin disease -

Exclusion Criteria:

History or presence of significant:

Cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrinal, immunologic, dermatologic, neurological or psychiatric disease.

More specifically, history or presence of significant:

Low birth weight babies (<2.5 Kg),

Malignancy,

Tuberculin positive,

Hodgkin's disease,

Corticosteroid therapy,

Generalised Eczema,

Infective dermatosis,

Hypogammaglobulinemia,

Immunosuppressed,

Above 14 years of age,

On anti-tubercular drugs,

Chest X ray evidence of TB.

-

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SR Lakshimipathy, MBBS, DCH, Principal Investigator — KC General Hospital, Malleswaram, Bangalore; Mohamed Kizhar Irshat, MBBS, DCH, Principal Investigator — Arya vysya maternity home & child welfare centre
Locations (1):
- Arya vysya maternity home & child welfare centre, Chennai, Tamil Nadu, India